CLINICAL TRIAL: NCT07254936
Title: The Comparison of Pain Using the Critical Care Pain Observation Tool Score With the Administration of Analgesic Doses of Ketamine and Dexmedetomidine in Post-Craniotomy Patients in the ICU
Brief Title: Comparison of Pain Using CPOT Score With Ketamine vs. Dexmedetomidine in Post-Craniotomy ICU Patients
Acronym: CPOT-KD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sumatera Utara (Other)
Responsible Party: Principal Investigator, Septani Anugrah Cinditya, Principal Investigator, Study Program Anesthesiology and Intensive Therapy, Universitas Sumatera Utara., Universitas Sumatera Utara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 50/KEPK/USU/2025; 50/KEPK/USU/2025 (Other: Universitas Sumatera Utara)
Record Dates: First submitted 2025-09-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Post-craniotomy Pain Management; Post-craniotomy; Pain Control in ICU; Ketamine vs Dexmedetomidine for Pain Relief
Keywords: CPOT; Post-craniotomy; Pain management; Ketamine; Dexmedetomidin; ICU pain control; Analgesics in ICU; Pain score assessment; Non-opioid analgesics
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a single-blind randomized controlled trial where participants are randomly assigned to one of two treatment groups. Group A will receive ketamine for pain management, while Group B will receive dexmedetomidine. Both groups will be evaluated for pain intensity using the Critical Care Pain Observation Tool (CPOT) at baseline, 6, 12, and 24 hours post-intervention. This parallel assignment design allows for a direct comparison of the effectiveness of these two analgesics in post-craniotomy ICU patients.
Who Masked: Participant
Masking Description: Masking Description:
  In this single-blind study, participants are blinded to the treatment they receive (ketamine vs. dexmedetomidine). The care providers and investigators are aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine for Pain Management (Other): This arm will receive ketamine as an analgesic to manage post-craniotomy pain in the ICU. Ketamine will be administered as an initial bolus dose of 0.2 mg/kg, followed by a continuous infusion of 0.1-0.2 mg/kg/h. Pain levels will be monitored using the Critical Care Pain Observation Tool (CPOT) at 6, 12, and 24 hours post-administration.
  Interventions: Drug: ketamine
- Dexmedetomidine for Pain Management (Other): This arm will receive dexmedetomidine as an analgesic to manage post-craniotomy pain in the ICU. Dexmedetomidine will be administered as an initial bolus dose of 1 mcg/kg, followed by a continuous infusion of 0.2-0.7 mcg/kg/h. Pain levels will be monitored using the Critical Care Pain Observation Tool (CPOT) at 6, 12, and 24 hours post-administration.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: ketamine — Ketamine will be administered as a bolus dose of 0.2 mg/kg, followed by a continuous infusion of 0.1-0.2 mg/kg/h for pain management in post-craniotomy ICU patients. Pain levels will be assessed using the Critical Care Pain Observation Tool (CPOT) at 6, 12, and 24 hours post-administration. This intervention aims to evaluate ketamine's effectiveness as an analgesic, providing pain relief while minimizing opioid usage.
  Arms: Ketamine for Pain Management
Drug: Dexmedetomidine — Dexmedetomidine will be administered as a bolus dose of 1 mcg/kg, followed by a continuous infusion of 0.2-0.7 mcg/kg/h for pain management in post-craniotomy ICU patients. Pain levels will be assessed using the Critical Care Pain Observation Tool (CPOT) at 6, 12, and 24 hours post-administration. This intervention aims to evaluate dexmedetomidine's effectiveness as an analgesic, offering sedation without respiratory depression.
  Arms: Dexmedetomidine for Pain Management

SUMMARY:
Study Overview:

This study is designed to compare two different medications used to manage pain after craniotomy surgery in the ICU. Craniotomy patients often experience severe pain, and it can be challenging to assess pain in patients who are unable to communicate. We are comparing the effectiveness of ketamine and dexmedetomidine in reducing pain, using the Critical Care Pain Observation Tool (CPOT) score to measure pain levels at different times after surgery.

Objective:

The goal is to determine which of these medications provides better pain relief for post-craniotomy patients in the ICU.

Study Design:

This study is a randomized controlled trial, meaning participants are randomly assigned to receive either ketamine or dexmedetomidine. The trial is single-blinded, which means the doctors administering the treatment will not know which medication the patient is receiving.

Why This Study is Important:

Managing pain effectively after surgery is crucial for recovery. Ketamine is known for its strong pain-relieving properties, while dexmedetomidine provides sedation without affecting breathing. This study will help doctors understand which medication is more effective in reducing pain for post-craniotomy patients.

DETAILED DESCRIPTION:
In this study, we will enroll post-craniotomy patients who are admitted to the ICU. They will be randomly assigned to one of two treatment groups: one group will receive ketamine, and the other will receive dexmedetomidine. Both groups will be given standard pain medication (ketorolac) along with their assigned intervention.

We will measure pain using the Critical Care Pain Observation Tool (CPOT), which evaluates pain based on observable signs such as facial expressions and body movements. CPOT scores will be recorded at several time points: 6 hours (T1), 12 hours (T2), and 24 hours (T3) after receiving the intervention.

Inclusion Criteria:

Patients over the age of 18

Post-craniotomy patients who are intubated and have a Glasgow Coma Scale (GCS) score between 8 and 15.

Exclusion Criteria:

Patients with hypersensitivity to ketamine or dexmedetomidine

Those with renal failure, heart failure, or hepatic failure

Patients who are unable to provide informed consent

Study Location:

This study will take place in the ICU of three hospitals in Medan: H. Adam Malik General Hospital, Hajj General Hospital, and TK II Putri Hijau Army Hospital.

Data Analysis:

After the data is collected, statistical tests will be conducted to determine whether ketamine or dexmedetomidine provides better pain relief. We will analyze CPOT scores from each group and compare the results at different time points (6, 12, and 24 hours).

This study aims to contribute valuable information to improve pain management strategies for post-craniotomy patients in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Intubated post-craniotomy patients in the ICU.
* Glasgow Coma Scale (GCS) score of 8-15 pre-operatively. Able to provide informed consent (either personally or through family/legal representative).

Exclusion Criteria:

* Hypersensitivity to ketamine or dexmedetomidine.
* Renal failure (elevated serum creatinine and BUN).
* Heart failure (EF <40%, elevated BNP/NT-proBNP, abnormal ECG).
* Hepatic failure (elevated AST/ALT, bilirubin, prolonged PT/INR).
* Patients with severe bradycardia, hypotension, or hallucinations due to study drugs.
* Death during the study period.
* New critical illness (e.g., sepsis, stroke).
* Withdrawal of consent by the patient or family.
* Incomplete data or ICU discharge before 24-hour follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (CPOT Score) | 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention.
  The Critical Care Pain Observation Tool (CPOT) will be used to assess pain intensity in post-craniotomy ICU patients.
  The CPOT scale ranges from 0 to 8, where higher scores indicate more severe pain.
  Pain assessments will be conducted at three time points: 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention.
  The primary outcome is the difference in mean CPOT scores between the ketamine and dexmedetomidine groups at each time point.

SECONDARY OUTCOMES:
Heart Rate Stability | Baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention
  Mean heart rate (beats per minute) will be recorded at baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention to evaluate cardiovascular stability between ketamine and dexmedetomidine groups.
Systolic Blood Pressure (SBP) Stability | Baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention
  Mean systolic blood pressure (mmHg) will be recorded at baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention to assess hemodynamic effects of ketamine and dexmedetomidine.
Diastolic Blood Pressure (DBP) Stability | Baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention
  Mean diastolic blood pressure (mmHg) will be recorded at baseline (T0), 6 hours (T1), 12 hours (T2), and 24 hours (T3) post-intervention to assess the effect of both drugs on vascular tone and perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- H. Adam Malik General Hospital, Hajj General Hospital, and TK II Putri Hijau Army Hospital, Medan, North Sumatra, Indonesia